CLINICAL TRIAL: NCT01544985
Title: A Randomized Double-blind Trial Comparing the Effect on Pain of an Oral Sucrose Solution Versus Placebo in Children 1 to 3 Months Old Needing Bladder Catheterization
Brief Title: Trial of an Oral Sucrose Solution Versus Placebo in Children 1 to 3 Months Old Needing Bladder Catheterization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Serge Gouin, Associate professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sucrose3456
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Pain
Keywords: pediatrics; emergency medicine; pain; bladder catheterization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sucrose po (Experimental): 88% sucrose solution (Syrup B.P.)
  Interventions: Drug: 88% sucrose po solution
- placebo po (Placebo Comparator): sterile water
  Interventions: Drug: placebo po

INTERVENTIONS:
Drug: 88% sucrose po solution — 88% sucrose solution (Syrup B.P.)
  Arms: sucrose po
Drug: placebo po — sterile water
  Arms: placebo po

SUMMARY:
INTRODUCTION AND JUSTIFICATION

The use of sucrose has been well studied for certain procedures in neonatal intensive care unit patients and in the newborn nursery settings, particularly for venous blood draws, capillary blood tests and circumcision. In these studies, infants receiving oral sucrose solutions before procedures cried less and had overall decreased behavioural pain responses when compared with those receiving placebo.

In Emergency Departments (ED), children undergo many painful procedures, such as bladder catheterization, capillary blood tests, venipuncture and lumbar puncture. Only two studies have examined the effectiveness of sweet solutions as an analgesic in the ED. A randomized controlled trial in an emergency setting of sucrose and/or pacifier for infants receiving venipuncture conducted by Curtis and al among infants of 0 to 6 months demonstrated a trend in reducing pain among the sub-group of infants of 0 to 3 months. However, this study showed no difference in pain scales after 3 months of age. Also, in a study examining the effect of sucrose during bladder catheterization, the subgroup of infants 1 to 30 days old who received a sweet solution showed smaller changes in pain scores, were less likely to cry during catheterization and returned to baseline more quickly, in comparison with the placebo group. However, among children of 31 to 90 days, there was no statistically significant difference in pain scores. In this study, they used a sucrose solution of only 24% and as they said in the discussion, it is possible that older infants, who on average received a smaller dose (in milligrams per kilogram), were in fact underdosed.

Finally, the painful procedure chosen for this study is bladder catheterization. Bladder catheterizations are frequently performed in the ED in this age group.

HYPOTHESIS The investigators believe that providing an oral sucrose solution during bladder catheterization will decrease pain levels in infants 1 to 3 months of age.

OBJECTIVES The investigators primary objective is to compare the efficacy an oral 88% sucrose solution to a placebo solution in reducing pain as assessed by the FLACC scale in children of 1 to 3 months during bladder catheterization in the ED. The investigators secondary objective is to asses changes in pain levels as per the NIPS score. The investigators will also measure variations in heart rate and crying time. All side effects will also be reported.

DETAILED DESCRIPTION:
INTRODUCTION AND JUSTIFICATION

Acute pain is one of the most common adverse stimuli experienced by children, occurring as a result of injury, illness, and necessary medical procedures. The American Academy of Pediatrics (AAP) and the American Pain Society (APS) have jointly issued a statement promoting the responsibility of paediatricians as leaders and advocates to ensure the humane and competent treatment of pain and suffering in all infants, children, and adolescents. Long-term effects of unmanaged pain in human infants have been shown to include permanent impairment of elements of cognitive development, such as learning, memory, and behaviour,and increased somatisation in childhood. The plasticity of the developing brain and the changes that occur in response to painful stimuli also contribute to altered perceptions of pain later in life. Early painful experiences affect children's future responses to analgesia. Weisman et al found that inadequate analgesia in young children during procedures diminished the effects of adequate analgesia during subsequent procedures. Many studies have suggested that the prompt and accurate recognition and treatment of pain in young infants is important for their immediate comfort and for their best possible lifelong development. Despite the recent interest in paediatric pain assessment, prevention and treatment, many children do not receive adequate management to alleviate pain. The ideal pre-procedural analgesic agent for minor invasive procedures would be a cost-effective, inexpensive, short-acting agent with few associated risks.

The use of sucrose has been well studied for certain procedures in neonatal intensive care unit patients and in the newborn nursery settings, particularly for venous blood draws, capillary blood tests and circumcision. In these studies, infants receiving oral sucrose solutions before procedures cried less and had overall decreased behavioural pain responses when compared with those receiving placebo. Furthermore, sucrose has been shown to be a safe intervention with no serious life-threatening adverse events and only few reported side effects consisting of minimal coughing with administration.

A Cochrane systematic review concluded that sucrose is safe and effective in reducing procedural pain from single short procedural events in neonates, but an optimal dose could not be identified due to inconsistency in effective sucrose dosage among studies. A review of published studies reported that sucrose or glucose in healthy term or preterm infants during single episodes of heel lancing, venipuncture or intramuscular injection is effective. However, uncertainties remain beyond the neonatal period, given the limited number of published studies.

In Emergency Departments (ED), children undergo many painful procedures, such as bladder catheterization, capillary blood tests, venipuncture and lumbar puncture. Only two studies have examined the effectiveness of sweet solutions as an analgesic in the ED. A randomized controlled trial in an emergency setting of sucrose and/or pacifier for infants receiving venipuncture conducted by Curtis and al among infants of 0 to 6 months demonstrated a trend in reducing pain among the sub-group of infants of 0 to 3 months. However, this study showed no difference in pain scales after 3 months of age. Also, in a study examining the effect of sucrose during bladder catheterization, the subgroup of infants 1 to 30 days old who received a sweet solution showed smaller changes in pain scores, were less likely to cry during catheterization and returned to baseline more quickly, in comparison with the placebo group. However, among children of 31 to 90 days, there was no statistically significant difference in pain scores. In this study, they used a sucrose solution of only 24% and as they said in the discussion, it is possible that older infants, who on average received a smaller dose (in milligrams per kilogram), were in fact underdosed. Moreover, they use the Douleur Aiguë du Nouveau-né (DAN) pain scale, which is less recognized than the FLACC scale to evaluate pain in such a study population. Finally, there were not enough participants between 30 and 90 days of age to obtain statistical significance for this age group.

Also, studies have used varieties of concentrations of sucrose (e.g. Rogers had used sucrose 24%, Curtis had used sucrose 44% and Lewindon had used sucrose 75%). Systematic reviews of the current literature have been unable to demonstrate superiority of one concentration of a sweet solution over another, but many studies suggest that higher concentrations of sweet solutions seem more effective. Therefore, the investigators chose to study the effect of a sweet solution named syrup B.P. (product by Laboratoire Atlas inc.) which contains 88% of sucrose. This solution is already commonly used in the population of infants up to 3 months of age and it is safe (e.g. prednisone syrup is made using this syrup). A 2 ml dose of 88% sucrose contains the same amount of carbohydrates as 25 ml of infant milk formulas which contain approximately 7,5g/100 ml. Also, 88% sucrose has the same concentration of sugar as many other medications which are commonly used in infants, such as oral antibiotics, oral steroid solutions and other pain medications. This syrup is of particular interest as it is of low cost ($9,58 for a bottle of 2000 ml), universally available, stable and viable for approximately three months. Therefore, the intervention studied here would be easy to apply in most clinical settings.

Finally, the painful procedure chosen for this study is bladder catheterization. Bladder catheterizations are frequently performed in the ED in this age group.

To date, there are no pain scales which have been validated precisely for the age group studied in this project. However, the Face, Legs, Activity, Cry and Consolability (FLACC) scale is recommended by the IMMPACT group (Initiative on Methods, Measurement and Pain Assessment in Clinical Trials). FLACC is an easily applicable pain scale in which the observer scores a patient on 5 categories, from 0 to 2 points, for a total score of maximum 10 points. The validity and reliability of this pain scale has been established in the past for children from 2 months to 7 years. Validity was evaluated by comparing the FLACC scale with the Objective Pain Scale and demonstrated that both tools showed similar behaviours (r=0.80; p<0.001). The interrater reliability between 2 observers was considered good (r[87]=0.94; p<0.001) with a kappa value greater than 0,50 for each category. Therefore, this pain scale was chosen as the measure of the investigators primary outcome, in this population of infants from 1 to 3 months old. Furthermore, the Neonatal Infant Pain Scale (NIPS) is a well validated pain scale for newborns up to 1 month of age. This pain scale was chosen as a secondary outcome. The investigators estimate that using one pain scale validated in infants up to 1 month of age and another validated in infants older than 2 months of age will allow us to assess pain in infants from 1 to 3 months of age best, given current available tools. Furthermore, other patient parameters such as heart rate and crying time will be used to corroborate findings.

HYPOTHESIS THe investigators believe that providing an oral sucrose solution during bladder catheterization will decrease pain levels in infants 1 to 3 months of age.

OBJECTIVES The investigators primary objective is to compare the efficacy an oral 88% sucrose solution to a placebo solution in reducing pain as assessed by the FLACC scale in children of 1 to 3 months during bladder catheterization in the ED. The investigators secondary objective is to asses changes in pain levels as per the NIPS score. The investigators will also measure variations in heart rate and crying time. All side effects will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Infants from 1 to 3 months (one month or more but less than 3 months old) of actual age (not corrected) requiring bladder catheterization as a part of their planned ED management while a research assistant is present.

Exclusion Criteria:

* Preterm infants (i.e. born <37 weeks)
* Urogenital anomalies
* Acute severe respiratory illness
* Chronic cardio-pulmonary condition
* Assisted ventilation (such as tracheostomy or oxygen dependance)
* Technology dependant (such as enteral feeding tube)
* Oropharyngeal malformation or dysfunction (such as cleft palate or micrognathia)
* Metabolic disease
* Previous participation in this study
* Painful procedures in the preceding 60 minutes (bladder catheterization, vesical puncture, lumbar puncture, capillary blood tests or IV insertion)
* Parental language barrier (French and/or English)

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Difference of pain scores using FLACC scale related to bladder catheterization | 1 minute

SECONDARY OUTCOMES:
Difference in pain scores using the NIPS scale related to bladder catheterization | 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Serge Gouin, MDCM, FRCPC, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Ste-Justine, Montreal, Quebec, Canada